CLINICAL TRIAL: NCT00551005
Title: Phase I Trial of Oral Etoposide in Combination With Celecoxib in Patients With Advanced Malignancies
Brief Title: Etoposide and Celecoxib in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 01036; P30CA033572 (NIH); CHNMC-01036; CDR0000570381 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-25; First posted 2007-10-30 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Celecoxib; Etoposide; Immunoenzyme Techniques

INTERVENTIONS:
Drug: celecoxib
Drug: etoposide
Other: immunoenzyme technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Etoposide and celecoxib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving more than 1 drug may be an effective treatment for advanced cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of celecoxib when given together with etoposide in treating patients with advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To describe the toxicities of the combination of oral etoposide at 50 mg daily with escalating doses of celecoxib in patients with advanced malignancies.
* To evaluate the effects of the combination of etoposide and celecoxib on plasma levels of vascular endothelial growth factor.

OUTLINE: This is a dose-escalation study of celecoxib.

In course 1, patients receive oral etoposide once daily on days 1-35 and oral celecoxib twice daily on days 8-35. In all subsequent courses, patients receive oral etoposide once daily and oral celecoxib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline, periodically during treatment, and at time of tumor progression. Samples are analyzed for vascular endothelial growth factor levels by enzyme-linked immunosorbent assay and stored for future analysis of circulating DNA of angiogenic biomarkers by polymerase chain reaction assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven diagnosis of a malignant disease for which no satisfactory treatment exists at the time of enrollment
* Patients with brain metastases which at the time of study enrollment are controlled and do not require treatment with corticosteroids are eligible

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* ANC > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L
* Creatinine clearance > 50 mL/min
* Serum bilirubin < 1.5 mg/dL
* AST and ALT < 2.0 times upper limit of normal (unless clearly due to the presence of tumor)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patient must be capable of understanding the nature of the trial and must give written informed consent

Exclusion criteria:

* Unstable or severe intercurrent medical conditions or active, uncontrolled infection
* History of allergic reactions to non-steroidal anti-inflammatory drugs (NSAIDs)
* History of bleeding peptic ulcer within the past 3 months

PRIOR CONCURRENT THERAPY:

Inclusion criteria:

* Recovered from all prior chemotherapy or radiotherapy
* Concurrent aspirin for cardiovascular indications allowed
* More than 2 weeks since prior and no other concurrent NSAIDs

Exclusion criteria:

* Had radiotherapy or chemotherapy within 3 weeks (nitrosoureas or mitomycin C within 6 weeks) prior to anticipated first day of dosing
* Undergoing concurrent therapy with other investigational agents or antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2001-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Toxicity
Maximum tolerated dose
Survival
Time to failure

CONTACTS AND LOCATIONS:
Overall Officials: Przemyslaw W. Twardowski, MD, Study Chair — City of Hope Comprehensive Cancer Center